CLINICAL TRIAL: NCT01187810
Title: A Phase I Study of Intravenous (Emulsion) Fenretinide (4-HPR, NSC 374551) in Children With Recurrent or Resistant Acute Lymphoblastic Leukemia (ALL), Acute Myelogenous Leukemia (AML), and Non-Hodgkin's Lymphoma (NHL) IND #70,058"
Brief Title: Fenretinide in Children With Recurrent/Resistant ALL, AML, and NHL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: drug supply
Sponsor: South Plains Oncology Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPOC2008-01
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma
Keywords: leukemia,lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Leukemia; Lymphoma | interventions — Fenretinide; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination of Fenretinide, Cytarabine, and Methotrexate (Experimental): IV for 7 days for each 21 day cycle
  Interventions: Drug: Fenretinide; Drug: Cytarabine; Drug: Methotrexate

INTERVENTIONS:
Drug: Fenretinide — 925 mg/m2 IV continuous infusion X 5 days for 6 cycles. Dose escalation will occur on a 3X3 basis.
  Other Names: N-(4-hydroxyphenyl) retinamide, 4-HPR
Drug: Cytarabine — dosing depending on age - will be administed intrathecally for all CNS negative subjects on day 0 and 15 of course 1, then on day 8 of each remaining cycle for CNS negative AML. For CNS positive ALL, NHL, and AML, will be administered alone on day 0 for and in combination with methotrexate and hydrocortisone on day 8, 15, 22 of cycle 1 and repeated on day 8 of each remaining cycle
  Other Names: Ara-C, Cytosine Arabinoside, Cytosar
Drug: Methotrexate — Dose depends on subject age - for CNS positive patients, will be given in combination with cytarabine and hydrocortisone on days 8, 15, and 22 during course 1. For courses 2-6, will be administered intrathecally on day 8 for CNS negative ALL and NHL. For patients who are CNS positive, it will be given in combination with cytarabine and hydrocortisone on day 8 of courses 2-6.
  Other Names: MTX, Amethopterin

SUMMARY:
The purposee of this study is to determine the safety and dosing of Fenretinide when given continuously for 5 days, every 3 weeks, in pediatric patients with recurrent and/or resistant acute lymphoblastic leukemia (ALL), acute myelogenous leukemia (AML), and non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
Fenretinide is a cytotoxic retinoid that has activity against a variety of cell lines in vitro in a dose-related manner. The exact mechanism of fenretinide cytotoxicity in leukemia and lymphoma cell lines is not known, but may include the de novo ceramide synthesis of ceramides and the generation of reactive oxygen species. The malignancy-specific nature of fenretinide-induced ceramides suggests that combinations of the drug with other ceramide modulating agents may have a favorable therapeutic index.

In this study, the primary aims are to define the maximum tolerated dose, toxicity profile, and pharmacokinetics of IV fenretinide when given continuously in pediatric patients with ALL, AML, and NHL. The drug will be administered via a central venous or percutaneous indwelling central catheter in an inpatient hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with relapsed or refractory ALL, AML, or NHL
* Must have had two or more therapeutic attempts for treating/curing disease
* Must have fully recoved from acute toxic effects of all prior therapy
* Karnofsky of greater than 50% for older than 10 years of age and Lansky greater than 50% for younger than 10 years.

Exclusion Criteria:

* Grade 2 Pruritus or Rash (all forms)
* Grade 3 Dry Skin that is refractory to topical medical management
* Cardiac Fractional Shortening < 27% on echocardiogram
* Left Ventricular Ejection Fraction < 45% on echocardiogram
* Known allergy to egg products or soy bean oil
* Renal, Liver, and Pancreatic function:

  * serum creatinine > 1.5X ULN
  * direct bilirubin > 1.5X ULN
  * ALT or AST > 2.5X ULN
  * Serum trigylcerides > 2.5X ULN for age
  * Lipase > 1.5X ULN for age
* History of pancreatitis

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2010-08; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose | end of study
Define systemic toxicities | end of study
Determine plasma pharmacokinetics | end of study

SECONDARY OUTCOMES:
Determine the response rate to IV Fenretinide | end of study
Determine bioavailability of fenretinide and metabolites | end of study
  To determine the bioavailability to cancer or peripheral blood mononuclear cells (PBMC) cells of fenretinide and metabolites delivered/obtained as an intravenous emulsion. To determine alterations to sphingolipid levels in PBMC and/or circulating leukemia blasts induced by fenretinide.

CONTACTS AND LOCATIONS:
Overall Officials: Anna R Franklin, MD, Study Chair — M.D. Anderson Cancer Center; Barry J Maurer, MD, PhD, Study Chair — Texas Tech University Health Sciences Center; Shengping Yang, PhD, Study Director — Texas Tech University Health Sciences Center; Min Kang, PharmD, Study Director — Texas Tech University Health Sciences Center; Patrick Reynolds, MD, PhD, Study Director — Texas Tech University Health Sciences Center
Locations (2):
- United States (2):
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided